CLINICAL TRIAL: NCT07369739
Title: Golidocitinib Combined With Selinexor for the Treatment of Chronic Active Epstein-Barr Virus Disease (CAEBVD): A Multicenter, Prospective, Single-arm Clinical Study
Brief Title: Golidocitinib Combined With Selinexor for CAEBVD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, doctor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS for CAEBVD
Record Dates: First submitted 2026-01-03; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lymphohistiocytosis; EBV; CAEBV
MeSH Terms: interventions — selinexor; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group:CAEBVD (Experimental)
  Interventions: Drug: golidocitinib; Drug: Selinexor (combination therapy)

INTERVENTIONS:
Drug: golidocitinib — golidocitinib 150 mg once daily.
Drug: Selinexor (combination therapy) — selinexor 40 mg once weekly.

SUMMARY:
This study is a multicenter, prospective, single-arm clinical investigation, with patients with CAEBVD as the main research subjects, to evaluate the effectiveness of the combined treatment regimen of golidocitinib and selinexor.

ELIGIBILITY:
Inclusion Criteria:

1. CAEBVD diagnosed in accordance with the Consensus on the Diagnosis and Treatment of Chronic Active Epstein-Barr Virus Disease (2025 Edition).
2. Aged ≥ 18 years and ≤ 70 years, regardless of gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Before the initiation of the study, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); total bilirubin ≤ 2 × ULN; serum creatinine ≤ 1.5 × ULN.
5. Routine blood test: absolute neutrophil count ≥ 1 × 10#/L; platelet count ≥ 50 × 10#/L; hemoglobin ≥ 60 g/L.
6. Coagulation function test requirements: international normalized ratio (INR) ≤ 2.0; prothrombin time (PT) ≤ 1.5 × ULN.
7. Women of childbearing potential must have a negative pregnancy test result, and be willing to take effective contraceptive measures during the trial period and for ≥ 12 months after the last dose; all male subjects must take contraceptive measures during the trial period and for ≥ 6 months after the last dose.
8. Signed informed consent form.

Exclusion Criteria:

1. Evidence of EBV-associated hematological diseases or malignancies, such as hemophagocytic lymphohistiocytosis, lymphomatoid granulomatosis, post-transplant lymphoproliferative disorder, non-Hodgkin's lymphoma, Burkitt lymphoma, nasopharyngeal carcinoma, and gastric cancer.
2. Having received any of the following treatments: prior treatment with any JAK inhibitor; administration of any investigational drug within 12 weeks prior to the first dose of the study drug; concurrent enrollment in another clinical study.
3. A history of other primary malignancies within 5 years prior to the first dose of the study drug, excluding locally curable malignancies that have received curative treatment (e.g., basal or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).
4. A history of organ transplantation (e.g., liver transplantation, kidney transplantation).
5. Planned hematopoietic stem cell transplantation during the study period.
6. Active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] at screening, or a peripheral blood hepatitis B virus DNA titer > 1×10³ copies/mL); active hepatitis C (defined as positive anti-hepatitis C virus antibody [HCV-Ab] and HCV-RNA at screening); positive serum HIV antigen or antibody; a history of syphilis.
7. Having undergone major surgery within 4 weeks prior to the first dose, or anticipating the need for major surgery during the study period.
8. Pregnant or lactating women.
9. A history of severe mental illness or drug abuse.
10. Uncontrolled infections (including pulmonary infection, intestinal infection); active major visceral hemorrhage (including gastrointestinal bleeding, alveolar hemorrhage, intracranial hemorrhage).
11. Hypersensitivity to the components of the study drug, or a history of severe allergic diathesis.
12. Patients who are unable to comply with the requirements during the trial and/or follow-up phase.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease Activity | Weeks 8 after the start of treatment
  Patients are classified into active and inactive phases based on their clinical symptoms, signs, and laboratory tests.Disease activity is defined as the presence of CAEBVD-related symptoms and signs.
EBV-DNA | Weeks 8 after the start of treatment
  The decline rate of EBV-DNA copy number in peripheral blood mononuclear cells (PBMCs)/plasma (defined as a 2-log reduction in EBV-DNA copy number) or conversion to negative.

OTHER OUTCOMES:
Survival | 6-month, 1-year and 2-year
  The 6-month, 1-year, and 2-year survival rates as well as the median survival time are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided